CLINICAL TRIAL: NCT06138951
Title: Dose Response Effect of Endurance Exercise on Protein Requirements of Endurance Athletes
Brief Title: Exercise Dose-response and Protein Requirements
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Daniel Moore, Associate Professor, University of Toronto
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: DRE
Record Dates: First submitted 2023-11-09; First posted 2023-11-18 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Exercise Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Nonexercised rested day (Placebo Comparator): Athlete will not exercise on trial day.
  Interventions: Other: Endurance exercise
- Recovery from 10KM run (Experimental): Athlete will run 10km on trial day.
  Interventions: Other: Endurance exercise
- Recovery from 20KM run (Experimental): Athlete will run 20km on trial day.
  Interventions: Other: Endurance exercise

INTERVENTIONS:
Other: Endurance exercise — On the trial day before commencing the indicator amino acid oxidation metabolic trial, participants will either rest, perform a 10km run on a treadmill, or perform a 20km run on a treadmill.

SUMMARY:
Study will investigate the impact of training volume on protein metabolism to estimate the impact on daily protein requirements of endurance athletes.

ELIGIBILITY:
Inclusion Criteria:

Healthy, male, endurance-trained participants who regularly run more than 40 km/week or perform endurance exercise for more than 4.5 hours/week

* Participants who have a self-reported 5-km run time of ≤23 min
* Participants who are categorized as at least "very good" based on a study by Shvartz & Reibold (Aviat Space Environ Med. 1990 Jan;61(1):3-11), in which VO2peak is used as an index. (i.e. the participants whose VO2peak is ≥57 ml/kg/min (18-24 y), ≥54 ml/kg/min (25-29 y), ≥52 ml/kg/min (30-34 y), ≥49 ml/kg/min (35-39 y)
* Ability to complete the 16-km familiarization run on Session 2
* Aged 18-40 years old

Exclusion Criteria:

* - Inability to meet health and physical activity guidelines according to the PAR-Q+.
* Female: hormonal fluctuations associated with the menstrual cycle have been reported to alter protein metabolism during exercise and may influence specific amino acid requirements at rest; as such, the present study will test the effect of endurance exercise on protein requirements in males only to ensure a stable hormonal environment and to increase the homogeneity of the physiological response. (NOTE: we plan to test females in a future trial based off of the results obtained herein)
* Inability to adhere to any of the protocol guidelines (i.e. alcohol, caffeine consumption)
* Regular tobacco use
* Illicit drug use (e.g. growth hormone, testosterone, etc.)

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2017-11-17 (Actual); Primary Completion 2018-08-15 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
Phenylalanine excretion | 8 hours
  Excretion of 13CO2 in the breath will be used to estimate the impact of exercise on daily protein requirements. This outcome will include the enrichment of 13CO2 in exhaled breath after the ingestion of [13C]phenylalanine tracer and the production of CO2 determined by indirect calorimetry at rest or after exercise.

SECONDARY OUTCOMES:
Phenylalanine flux | 8 hours
  The enrichment of [13C]phenylalanine in the urine will be used to estimate the flux of phenylalanine in the body at rest or after exercise.
Phenylalanine oxidation | 8 hours
  The oxidation of [13C]phenylalanine will be determined by correcting phenylalanine excretion by phenylalanine flux.

CONTACTS AND LOCATIONS:
Locations (1):
- Goldring Centre for High Performance Sport at the University of Toronto, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No